CLINICAL TRIAL: NCT07204392
Title: Unveiling the Germline Predisposition to Myeloproliferative Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Elisa Rumi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: U27_MPN
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Myeloproliferative Disease; Germline Mutation
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The classic Ph-negative myeloproliferative neoplasms (MPN) are a group of clonal hematopoietic disorders caused by a dysregulated JAK/STAT signal transduction because of acquired somatic mutations of JAK2, CALR or MPL genes. They are sporadic diseases but there are several lines of evidence that support the role of germline factors in the pathogenesis of MPN: the existence of familial clustering, the presence of more than one clone in some patients, the known existence of common polymorphisms that cause predisposition to MPN.

In this study, we would like to define the germline predisposition to MPN.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PV, ET, prePMF, overt PMF or MPN-U according to 2016 WHO criteria
* Characterization of the MPN driver mutation performed at any moment before enrolment
* diagnosis of MPN made when the patient was younger than 27 years old OR at least a second case of hematologic malignancies in first or second-degree relatives

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected with early-onset or familial myeloproliferative
Sampling Method: Non-Probability Sample
Enrollment: 313 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify a germline predisposition to MPN through the application of an NGS-based gene panel test in young patients. | 3 years
To identify the germline genetic factors that underlie familial clustering of MPN through whole genome sequencing (WGS). | 3 years

SECONDARY OUTCOMES:
To identify phenotype-genotype correlations: we aim to correlate the molecular data with clinical data and relevant outcomes | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No